CLINICAL TRIAL: NCT07076576
Title: The Investigation the Effects of Yoga on Attention,Hyperactivity- Impulsivity and Motor Skills in Children With Attention Deficit Hyperactivity Disorder
Brief Title: Effects of Yoga in Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Elif Nur Taşcıoğlu, Research Assistant, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAU-FTR-ENT-001
Record Dates: First submitted 2025-03-07; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD); Yoga; Motor Skills
Keywords: Attention Deficit Hyperactivity Disorder; Yoga; Motor Skills
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga Training (Experimental): The children in the experimental group underwent yoga training.
  Interventions: Other: Yoga Training
- Control Group (No Intervention): The participants in the control group continued to their medication treatment and have not received any additional intervention.

INTERVENTIONS:
Other: Yoga Training — The children in the experimental group underwent yoga training for a total of 16 sessions consisting of 45 minutes each session, 2 times a week for 8 weeks.
  Arms: Yoga Training

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is characterized by symptoms of inattention, impulsivity, and hyperactivity. Due to the core symptoms of ADHD, more than 30-50% of children with the disorder may experience impaired motor abilities.

The aim of this study is to investigate the effects of yoga on core ADHD symptoms and motor skills. Thirty-three children with ADHD (ages 6-12) who are undergoing medication were randomly divided into two groups. The intervention group will participate in yoga sessions twice a week for 8 weeks, while the control group will not receive any additional intervention.

The Turgay Disruptive Behavior Disorders Rating Scale will be used to assess ADHD symptoms, and Cognitive Disengagement Syndrome will be evaluated using the Children and Adolescent Behavior Inventory (CABI) Family Questionnaire by a child and adolescent psychiatrist. Additionally, the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition-Short Form, will be administered by a physiotherapist to assess motor skills before, after, and one month following the intervention.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is a neurodevelopmental disorder characterized by symptoms of inattention, impulsivity, and hyperactivity. Due to these core symptoms, more than 30-50% of children with ADHD may experience impaired motor abilities.

Symptoms of ADHD include difficulty maintaining focus on tasks for extended periods, forgetfulness, restlessness, fidgeting, impatience, trouble waiting in line, frequent interruptions, frequent falls, injuries, and clumsiness. Additionally, 39% of children with ADHD also have Cognitive Disengagement Syndrome (CDS), which is characterized by symptoms such as daydreaming, slow and limited movement, appearing drowsy and lethargic, blank staring, looking confused, and impairments in motor and cognitive skills. CDS has been linked to psychopathology and functional impairments, including symptoms of depression and anxiety, independent of ADHD.

Treatment options for ADHD include both pharmacological and nonpharmacological approaches. Due to its neurological basis, pharmacological treatments are typically the first-line intervention. However, physical exercise interventions such as yoga are also considered alternative therapeutic options. Yoga requires participants to perform complex motor skill combinations accurately and fluidly. Research suggests that yoga enhances dopamine and serotonin levels, which play a role in modulating motor, executive, impulsive, and cognitive functions. As a mind-body intervention, yoga improves attention and inhibitory control, making it an enjoyable and effective therapeutic approach for children with attention deficits. The aim of our study was to examine the effects of an 8-week yoga intervention on core symptoms, Cognitive Disengagement Syndrome, and motor skills in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 12 years
* Able to understand and accept verbal instructions
* Using medication which includes methylphenidate
* After the titration period, the drug dose should be between 0.6-1 mg/kg
* Not participating in any additional intervention programs other than the medication treatment initiated after the diagnosis
* The child and the parent being willing to participate in the study

Exclusion Criteria:

* Having comorbid diagnoses such as specific learning disorder, autism spectrum disorder, psychotic disorder, bipolar disorder, or mental retardation
* Having a neurological, metabolic, or orthopedic condition such as head trauma, cerebral palsy, epileptic seizures, or visual and speech impairments.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
ADHD Symptoms | Baseline (pre-intervention), post-intervention (after 8 weeks of intervention for the Yoga group or 8 weeks after baseline for the Control group), and at 1-month follow-up (1 month after post-intervention assessment)
  The Turgay ADHD Scale will be used to assess ADHD symptoms administered by parents. The scale has been developed by Turgay to assess disruptive behavior disorders with DSM IV diagnostic criteria. The The scale has 41 items: 9 for attention deficit, 6 for hyperactivity, 3 for impulsivity, 8 for oppositional defiant disorder, and 15 for conduct disorder.
Motor Skills | Baseline (pre-intervention), post-intervention (after 8 weeks of intervention for the Yoga group or 8 weeks after baseline for the Control group), and at 1-month follow-up (1 month after post-intervention assessment)
  A pediatric physiotherapist will be used to assess motor skills with the Bruininks-Oseretsky Test of Motor Proficiency Test-Short Form (BOT2-SF) before, after, and one month after treatment. The Bruininks-Oseretsky Test of Motor Proficiency is used to assess the motor competence of children and adolescents between the ages of 4 and 21. The test's short form, BOT2-SF, is constructed of eight subtests totaling 12 items. The subtests are as follows: fine motor precision, fine motor integration, manual skills, bilateral coordination, balance, speed and agility, upper extremity coordination, endurance.

SECONDARY OUTCOMES:
Cognitive Disengagement Syndrome (Sluggish Cognitive Tempo) | Baseline (pre-intervention), post-intervention (after 8 weeks of intervention for the Yoga group or 8 weeks after baseline for the Control group), and at 1-month follow-up (1 month after post-intervention assessment)
  Cognitive Disengagement Syndrome was evaluated using a Children and Adolescent Behavior Inventory (CABI) Family Questionnaire administered by parents. This scale asks parents and caregivers about their child's or adolescent's behavior. It consists of nine subscales and 67 items, each of which can be used independently. The first subscale, comprising 15 items, evaluates SCT. Responses are rated on a 6-point Likert scale, ranging from 0 (almost never) to 5 (almost always).
Clinical Global Impressions - CGI | Baseline (pre-intervention), post-intervention (after 8 weeks of intervention for the Yoga group or 8 weeks after baseline for the Control group), and at 1-month follow-up (1 month after post-intervention assessment)
  The Clinical Global Impressions (CGI) Scale will be administered by parents. This assessment is a standardized measure used by clinicians to rate disease severity, changes over time, and the effectiveness of treatment. It consists of three subscales. The first subscale is ''Severity of Illness'' and the second subscale is ''Clinical Global Impression Improvement'' will be used in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No